CLINICAL TRIAL: NCT04177862
Title: Sublingual Sufentanil vs Intravenous Fentanyl for Acute Pain in the Ambulatory Surgery Center
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES-2019-28303
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pain; Pain, Acute; Anesthesia
MeSH Terms: conditions — Pain; Acute Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Sufentanil (Experimental): Single dose of sublingual sufentanil for acute pain.
  Interventions: Drug: Sublingual Sufentanil
- IV Fentanyl (Active Comparator): single dose of IV fentanyl for acute pain.
  Interventions: Drug: IV Fentanyl

INTERVENTIONS:
Drug: Sublingual Sufentanil — 30 mcg of sublingual sufentanil
  Arms: Sublingual Sufentanil
Drug: IV Fentanyl — 50 mcg of IV fentanyl
  Arms: IV Fentanyl

SUMMARY:
The purpose of this study is to determine if a single dose of sublingual sufentanil is as or more efficacious than a single dose of IV fentanyl in a post anesthesia care setting.

DETAILED DESCRIPTION:
This is a level I randomized prospective outcomes study comparing two groups of patients. Upon arrival in the ambulatory surgery center (ASC) post-anesthesia care unit (PACU) if the patient has a pain score of 4 or greater they will then be randomized to one of two groups. Group 1 will receive 50 mcg of IV fentanyl and group 2 will receive 30 mcg of sublingual sufentanil. The primary outcome assessed will be time of readiness to discharge after arrival in the post-anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* undergoing outpatient ambulatory surgery
* recipient of general anesthesia
* pain score of 4 or greater in the PACU

Exclusion Criteria:

* non-english speaking patients
* cancer surgeries
* patients who have allergy or intolerance to the study drugs or derivatives
* patients on chronic opioids (defined as daily opioids for 3 months or longer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Berg, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to groups after undergoing their surgical procedures if they had a self-reported pain score of 4 and above on the 11-point numeric rating scale during phase 1 of PACU.
Groups:
- Sublingual Sufentanil: Single dose of sublingual sufentanil for acute pain.
  Sublingual Sufentanil: 30 mcg sublingual sufentanil tablet
Period: Overall Study
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Started (Allocated to intervention) | 35 | 40
Completed | 33 | 33
Not Completed | 2 | 7
Not completed — Protocol Violation | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Sufentanil | IV Fentanyl | Total
Number analyzed (Participants) | 35 | 40 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [32.5 to 58] | 37 [22.75 to 53.75] | 42 [25.5 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 40 | 75

OUTCOME MEASURES:

1. Primary Outcome: Recovery Room Time
Description: The time (reported in minutes) from when the patient arrives in the PACU, right after surgery, to the time that all discharge criteria are met.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
minutes | 73.0 [56.0 to 89.0] | 65.0 [56.0 to 89.0]

2. Secondary Outcome: Rescue Milligram Morphine Equivalents (Opioid Use After Intervention Until Discharge)
Description: All doses of opioid medications administered following initial dosage (sufentanil or fentanyl depending on study arm) will be converted to milligram morphine equivalents and summed for reporting.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
milligram morphine equivalents | 15.0 [7.5 to 30.0] | 22.5 [13.1 to 23.4]

3. Secondary Outcome: Adverse Events
Description: Number of serious adverse events (grades 3, 4, and 5) experienced by each group
Time Frame: 1 day
Measure: Number; unit: SAEs
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
SAEs | 0 | 0

4. Secondary Outcome: Postoperative Nausea and Vomiting (PONV)
Description: Number of participants in each arm who are treated for nausea and/or vomiting.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
Participants | 4 | 7

5. Secondary Outcome: Supplemental Oxygen
Description: Number of participants in each arm who require supplemental oxygen therapy
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
Participants | 4 | 4

6. Secondary Outcome: Overall Benefit of Analgesic Score (OBAS)
Description: Overall Benefit of Analgesic Score (OBAS) is a 7-item multi-dimensional survey that assesses analgesia benefits. Items are scored on a scale from 0 (minimal) to 4 (maximal). Total score is a sum of the 7 item scores with question 7 scored as 4 minus the patient reported number. Total scores range from 0 to 28 with lower scores representing greater benefit from analgesic therapy.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sublingual Sufentanil | IV Fentanyl
Number analyzed (Participants) | 35 | 40
score on a scale | 3.0 [2.0 to 4.0] | 3.0 [1.0 to 4.5]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Sublingual Sufentanil | IV Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/40
Other Adverse Events (participants affected / at risk) | 4/35 | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual Sufentanil (N=35) | IV Fentanyl (N=40)
Postoperative nausea (Surgical and medical procedures) | 4 (4) | 7 (7) — Postoperative nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT04177862/Prot_SAP_000.pdf